CLINICAL TRIAL: NCT03915262
Title: Exocrine Pancreatic Insufficiency's Prevalence in Active Crohn's Disease Treated by Biological Therapy
Brief Title: Exocrine Pancreatic Insufficiency's Prevalence in Active Crohn's Disease
Acronym: IPEC
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0294
Record Dates: First submitted 2019-04-09; First posted 2019-04-16 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn's Disease
  Interventions: Biological: Search for exocrine pancreatic insufficiency at week 0 and 12

INTERVENTIONS:
Biological: Search for exocrine pancreatic insufficiency at week 0 and 12 — We will collect 24 hours stool to search for steatorrhea, and to measure elastase and calprotectin.
  We will collect a total of 8 additional blood tubes (25mL), during regular blood sampling for a patient under biological therapy for a Crohn's disease.
  We will gather the total caloric and fat intake with a diet record.

SUMMARY:
This study aims to assess the prevalence of exocrine pancreatic insufficiency (EPI) in a population of patients with active Crohn's disease. Studies already describe a prevalence rate around 18-66%. In this multicentric prospective study, we plan to compare EPI's prevalence at week 0 and week 14 of an induction phase of a biological therapy. The biological therapy will be initiate for an active Crohn's disease. Secondary outcomes will be: malnutrition's prevalence, and Crohn's disease activity level.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or more
* Crohn's disease diagnosed for more than 3 months.
* Active Crohn's disease : CDAI score > 150 + [CRP > 5 mg/L or faecal calprotectin > 250mcg/g or endoscopic lesion or MRI lesion]
* Indication of a biological therapy (anti-TNFα, vedolizumab ou ustekinumab).

Exclusion Criteria:

* Crohn's disease that doesn't fit the previous criteria
* Extended resection of small intestine (>40cm)
* Chronic pancreatitis diagnosed before inclusion
* Contraindication to biological therapy (anti-TNFα, vedolizumab ou ustekinumab)
* Pancreatic enzyme replacement therapy
* Pregnant or breastfeeding woman
* Patient under the protection of a conservator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an active Crohn's Disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-11-15 (Actual); Primary Completion 2026-11-15 (Estimated); Study Completion 2027-11-15 (Estimated)

PRIMARY OUTCOMES:
Exocrine pancreatic insufficiency's prevalence | week 0
  Exocrine pancreatic insufficiency will be defined as the association of : fecal elastase <200 mcg/g and steatorrhea (>7g of fecal fat per day) or an fat absorption rate < 95%
Exocrine pancreatic insufficiency's prevalence | week 14
  Exocrine pancreatic insufficiency will be defined as the association of : fecal elastase <200 mcg/g and steatorrhea (>7g of fecal fat per day) or an fat absorption rate < 95%

CONTACTS AND LOCATIONS:
Overall Officials: Gilles BOSCHETTI, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Service d'Hépato-Gastroentérologie, Centre Hospitalier Lyon-Sud, HCL, Pierre-Bénite, France

IPD SHARING:
Plan to Share IPD: Undecided